CLINICAL TRIAL: NCT06630572
Title: Rifaximin Blunted Higher Levels of Endotoxin in Cirrhosis Patients: a Randomized, Double Blind, Short Term Interventional Trial
Brief Title: Rifaximin in Cirrhosis: Effects on Endotoxin and Haemostatic Indexes
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Because drug is expired
Sponsor: University of Roma La Sapienza (Other)
Collaborators: Azienda Policlinico Umberto I (Other)
Responsible Party: Principal Investigator, Stefania Basili, Clinical Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT 2017-000488-34
Record Dates: First submitted 2018-01-18; First posted 2024-10-08 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-08

CONDITIONS: Liver Cirrhosis; Coagulation Disorder; Platelet Disorder; Endotoxemia
Keywords: Rifaximin; Liver Cirrhosis; Endotoxin; Platelet function
MeSH Terms: conditions — Liver Cirrhosis; Hemostatic Disorders; Blood Platelet Disorders; Endotoxemia | interventions — Rifaximin

STUDY DESIGN:
Intervention Model Description: Randomized, placebo control, double-blind trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TREATMENT (Experimental): Rifaximin (1100 mg/die) - 550 b.i.d.
  Interventions: Drug: Rifaximin
- PLACEBO (Placebo Comparator): Placebo - b.i.d.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rifaximin — Patients randomized to receive Rifaximin for 14 days
  Arms: TREATMENT
Drug: Placebo — Patients randomized to receive Placebo for 14 days
  Arms: PLACEBO

SUMMARY:
Rifaximin is an antibiotic that acts locally in the gastrointestinal tract with a broad spectrum of antibacterial activity. The efficacy of rifaximin is well documented in the prevention of acute hepatic encephalopathy. There is no evidence on its benefit to modulate hypercoagulative state in cirrhotic patient.

To assess the effect of a short-term treatment with rifaximin on systemic levels of intestinal endotoxin and on platelet and coagulation markers in patients with decompensated cirrhosis the study has been planned.

DETAILED DESCRIPTION:
The term coagulopathy has been coined because of impaired clotting activation detected by laboratory tests in association with deterioration of liver function; the frequent coexistence of hyperfibrinolysis, low platelet count, and platelet dysfunction reinforced the concept that coagulopathy is associated with cirrhosis.

This concept has been recently challenged for several reasons. The prolongation of global tests of clotting activation does not actually reflect hemostatic changes in vivo and maybe a laboratory artefact. In addition, cirrhotic patients actually disclose a tendency to a hypercoagulation state, which seems to be related to endotoxemia and may be detected in both peripheral and portal circulation, and to an increased platelet activation.

Bacterial lipopolysaccharide (LPS, endotoxin) is elevated in cirrhosis, particularly in decompensated cirrhosis, with a mechanism related to an enhanced gut permeability and ensuing translocation of LPS in the peripheral circulation. Recent data demonstrated that cirrhosis is associated with a low-grade endotoxemia, which is more evident in Child-Pugh classes B and C. Of note, LPS significantly correlated with sCD40L and sPs, suggesting a role for LPS in eliciting platelet activation.

It is difficult to believe that under these circumstances patients with cirrhosis are at high risk of bleeding; thus, apart from gastrointestinal tract bleeding, which is independent of changes of the clotting system, spontaneous bleeding in cirrhosis is rare. Conversely, in vivo data reporting the existence of platelet and clotting activation may explain the increased risk for thrombosis overall in portal circulation. This opens a new and interesting scenario as portal vein thrombosis, which may occur in approximately 20% of cirrhotic patients, should be treated with antithrombotic drugs (https://clinicaltrials.gov/ct2/show/NCT01470547). However, planning trials with anticoagulants in cirrhosis will be very difficult because the persistent concept of "coagulopathy in cirrhosis" is likely to be a barrier against the use of anticoagulants.

Interventional trials to modulate low-grade endotoxemia are warranted to assess if this therapeutic approach may reduce the risk of thrombosis in cirrhosis.

In a small cohort of cirrhotic, a previous study demonstrated that administration of non-absorbable antibiotic reduces thrombin generation coincidentally with serum LPS reduction suggesting a role for LPS as trigger of clotting activation. No data were provided, however, on the effect of this treatment on platelet activation or on the duration of clotting system inhibition.

Rifaximin is an antibiotic that acts locally in the gastrointestinal tract with a broad spectrum of antibacterial activity. The efficacy of rifaximin is well documented in the prevention of acute hepatic encephalopathy (HE). It is recommended as a first-line therapy for HE and was recently approved for the prevention of HE in high-risk populations. More recently, clinical trials have been performed to evaluate the effect of this drug on the prophylaxis of spontaneous bacterial peritonitis (SBP) and other cirrhosis-related complications. Although these studies demonstrated excellent prospects for the clinical application of rifaximin, there is no evidence on its benefit to modulate hypercoagulative state in the cirrhotic patient.

Study objective: to assess the effect of a short-term (14 days) treatment with rifaximin (1100 mg/die) on systemic levels of intestinal endotoxin and on platelet and coagulation markers in patients with decompensated cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years
* Patients of Child-Pugh grade B or C (decompensated liver cirrhosis, as confirmed by clinical symptoms and signs, laboratory results, ultrasound and spiral computed tomography)

Exclusion Criteria:

* Presence of overt infection or sepsis
* Treatment with systemic or non-absorbable antibiotic, aspirin or other non-steroidal anti-inflammatory drugs, antidepressant drugs in the previous 30 days
* Recent need of transfusion of platelets or plasma
* Presence of extra-hepatic malignancy
* Active alcohol intake in the last 6 months
* Pregnancy or breast feeding
* Presence of overt HE, GI haemorrhage, SBP or other concurrent infections during the previous one month
* Human immunodeficiency virus (HIV) infection
* Chronic renal and/or respiratory insufficiency
* Severe heart disease
* Allergy to rifaximin
* Active post-viral hepatitis requiring or on direct-acting antiviral (DAA) agents
* Previous or active intestinal obstruction.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-04-03 (Actual); Primary Completion 2022-04-03 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Decrease in serum endotoxemia after 14-day treatment with Rifaximin. | 14, 30, 60 Days
  Significant decrease (-20%) in serum bacterial LPS (endotoxemia) after 14-day treatment with Rifaximin 550 mg b.i.d respect to the control group as well as after 30 and 60 days from the end of the treatment.

SECONDARY OUTCOMES:
Impact of serum changes of LPS on coagulation and/or platelet indexes | 14, 30, 60 Days
  Significant correlation between change in serum LPS and thrombin generation and/or platelet activation indexes in both groups to support the role of LPS as trigger of clotting activation and platelet activation.
Clinical Failure | 14, 30, 60 Days
  Proportion of patients with clinical failure.
Safety and tolerability: Number of participants with adverse events as a measure of safety and tolerability | 14, 30, 60 Days
  Number of participants with adverse events as a measure of safety and tolerability

OTHER OUTCOMES:
Platelet activation | 14, 30, 60 Days
  Evaluation of soluble markers of platelet activation [Flow cytometric analysis and ELISA]
Platelet- leukocyte aggregation | 14, 30, 60 Days
  Evaluation of platelet-leukocyte aggregates by Flow cytometric analysis
Platelet turnover | 14, 30, 60 Days
  Determination of platelet indices indicative of elevated platelet turnover.
Gut microbiota | 14, 30, 60 Days
  Evaluation of intestinal barrier permeability, by ELISA for LPS, marker of gut permeability.
Neutrophil extracellular traps (NETs) | 14, 30, 60 Days
  Soluble markers of neutrophil extracellular trap (NET) in circulation.
Gut microbiota | 14, 30, 60 Days
  Evaluation of intestinal barrier permeability, by ELISA for Zonulin, marker of gut permeability.

CONTACTS AND LOCATIONS:
Overall Officials: Stefania BASILI, Prof., Study Chair — SAPIENZA UNIVERSITY- Department of Translational and Precision Medicine; Oliviero Riggio, Prof., Principal Investigator — SAPIENZA UNIVERSITY- Department of Translational and Precision Medicine; Manuela Merli, Prof., Principal Investigator — SAPIENZA UNIVERSITY- Department of Translational and Precision Medicine; Lucia Stefanini, Prof., Principal Investigator — SAPIENZA UNIVERSITY- Department of Translational and Precision Medicine; Roberto Carnevale, Prof., Principal Investigator — SAPIENZA UNIVERSITY
Locations (1):
- Sapienza University of Rome - Policlinico Umberto I Roma, Rome, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Violi F, Ferro D. Clotting activation and hyperfibrinolysis in cirrhosis: implication for bleeding and thrombosis. Semin Thromb Hemost. 2013 Jun;39(4):426-33. doi: 10.1055/s-0033-1334144. Epub 2013 Mar 13. PMID 23487343
- [Background] Violi F, Ferro D, Basili S, Lionetti R, Rossi E, Merli M, Riggio O, Bezzi M, Capocaccia L. Ongoing prothrombotic state in the portal circulation of cirrhotic patients. Thromb Haemost. 1997 Jan;77(1):44-7. PMID 9031447
- [Background] Nolan JP. The role of intestinal endotoxin in liver injury: a long and evolving history. Hepatology. 2010 Nov;52(5):1829-35. doi: 10.1002/hep.23917. PMID 20890945
- [Background] Raparelli V, Basili S, Carnevale R, Napoleone L, Del Ben M, Nocella C, Bartimoccia S, Lucidi C, Talerico G, Riggio O, Violi F. Low-grade endotoxemia and platelet activation in cirrhosis. Hepatology. 2017 Feb;65(2):571-581. doi: 10.1002/hep.28853. Epub 2016 Nov 5. PMID 27641757
- [Background] Violi F, Basili S, Raparelli V, Chowdary P, Gatt A, Burroughs AK. Patients with liver cirrhosis suffer from primary haemostatic defects? Fact or fiction? J Hepatol. 2011 Dec;55(6):1415-27. doi: 10.1016/j.jhep.2011.06.008. Epub 2011 Jun 28. PMID 21718668
- [Background] Ferro D, Angelico F, Caldwell SH, Violi F. Bleeding and thrombosis in cirrhotic patients: what really matters? Dig Liver Dis. 2012 Apr;44(4):275-9. doi: 10.1016/j.dld.2011.10.016. Epub 2011 Nov 25. PMID 22119620
- [Background] Bass NM, Mullen KD, Sanyal A, Poordad F, Neff G, Leevy CB, Sigal S, Sheikh MY, Beavers K, Frederick T, Teperman L, Hillebrand D, Huang S, Merchant K, Shaw A, Bortey E, Forbes WP. Rifaximin treatment in hepatic encephalopathy. N Engl J Med. 2010 Mar 25;362(12):1071-81. doi: 10.1056/NEJMoa0907893. PMID 20335583
- [Background] Rivkin A, Gim S. Rifaximin: new therapeutic indication and future directions. Clin Ther. 2011 Jul;33(7):812-27. doi: 10.1016/j.clinthera.2011.06.007. Epub 2011 Jul 7. PMID 21741091
- [Background] Danulescu RM, Ciobica A, Stanciu C, Trifan A. The role of rifaximine in the prevention of the spontaneous bacterial peritonitis. Rev Med Chir Soc Med Nat Iasi. 2013 Apr-Jun;117(2):315-20. PMID 24340510